CLINICAL TRIAL: NCT07402109
Title: Organ Sparing Marker-less CBCT-guided Stereotactic Adaptive Radiotherapy for Primary Non-metastasized Renal Tumors
Brief Title: CBCT Guided Markerless SBRT for Renal Cell Cancer
Acronym: CT-STARRS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, E. (Euphemia) A.M. Froklage, Radiation Oncologist, MD PhD, principal investigator, Erasmus Medical Center
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NL-010279
Record Dates: First submitted 2025-09-30; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Renal Cell Carcinoma (RCC)
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Additional imaging (Experimental): Additional CBCT scans will be made after each fraction, follow-up will be done using photon counting CT
  Interventions: Radiation: Additional radiation due to imaging

INTERVENTIONS:
Radiation: Additional radiation due to imaging — Additional imaging will be done using CT, therefore the patient will receive additional radiation dose

SUMMARY:
This study aims to improve the treatment of kidney tumors using radiotherapy, by investigating whether kidney cancer can be more effectively irradiated with the help of new imaging techniques

DETAILED DESCRIPTION:
In total 40 patients will be treated for RCC using SBRT.

For 15 patients, additional breath-hold CBCT scans will be made during SBRT to investigate the intra- and inter-fraction uncertainty in breath-hold positions as well as assessing the feasibility of using surface guidance as a surrogate for target position.

Subsequently, 25 patients will be treated using the new motion management technique developed using the extra imaging data obtained from the first cohort of patients. It is hypothesized that either breath-hold or gating in combination with surface guidance will result in a reproducible (stable) position of the target and therefore minimal margins.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven non-metastastic RCC or high suspicion of RCC based on imaging without histological evidence
* No metastatic lesions
* Patients must be 18 years or older
* Ability to understand the requirements of the study and to give written informed consent, as determined by the treating physician.

Written informed consent

Exclusion Criteria:

* Previous high-dose radiotherapy in the region of the kidney

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Reduction of renal dose | At day 1 planning CTs are acquired for treatment planning. These scans will be used to make a treatment planning with standard motion management and a treatment planning will be made using novel motion management. Both plans will be compared.
  The primary aim of this project is to minimize treatment margins, reducing the PTV, to optimally preserve renal function, while ensuring adequate tumor coverage as well as adhering to dose constraints of OARs. Primary endpoint of this study is the reduction of dose to the healthy ipsilateral kidney, defined as the ipsilateral renal volume receiving 50% of the prescribed dose (V50%).

SECONDARY OUTCOMES:
Evaluate the current treatment, including the benefit of online adaptive radiotherapy | Day 1 planning CTs. Approximately day 14: start radiotherapy (3 times per week). At each fraction: CBCT. At completion of treatment (at approximately day 30) planning for adapted and non-adapted plans
  The possible benefit of online adaptive radiotherapy will be assessed by doing an offline analysis by comparing target coverage in % between adapted and non-adapted, original plans
Investigate treatment fraction reduction | At day 1 planning CTs are acquired for treatment planning. These will be used for treatment planning for simulated fraction schedules using standard and novel motion management
  the feasibility of transitioning from a 5×8 Gy schedule to 3×14 Gy or 1×26 Gy will be investigated by simulating the difference in the mean number of fractions when using SoC motion management and the novel motion management
Change From Baseline in Tumor Contrast Enhancement on Photon-Counting CT | Baseline (pre-treatment) and follow-up at 3, 6, and 12 months after completion of treatment
  Tumor contrast enhancement measured on contrast-enhanced photon-counting CT scans. Enhancement values will be quantified within the treated lesion and reported as change from baseline.
Change From Baseline in Tumor Iodine Concentration on Photon-Counting CT | Baseline (pre-treatment) and follow-up at 3, 6, and 12 months after completion of treatment
  Iodine concentration quantified within the treated lesion using material decomposition from contrast-enhanced photon-counting CT scans. Values will be reported as change from baseline.

OTHER OUTCOMES:
Monitor side effects | During treatment and at 3, 6, and 12 months after completion of treatment
  Side-effects are assessed during treatment and follow up, according to Common Terminology Criteria for Adverse Events version 5 (CTC-AE version 5).
Monitor renal function | At 3, 6, and 12 months after treatment, followed by biannual evaluations at the referring center (referring urologist) in the second year and annual assessments in the third and fourth years
  Renal function changes will be measured using estimated glomerular filtration rate (eGFR)